CLINICAL TRIAL: NCT02830490
Title: Test-retest Reliability and Minimal Detectable Change Scores for the Short Physical Performance Battery (SPPB), One Leg Balance and Timed up and go.
Brief Title: Reliability of Functional Measures in Hemodialysis Patient.
Status: Completed | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Eva Segura Ortí, PhD, Cardenal Herrera University
Other Study IDs: CardenalHU
Record Dates: First submitted 2015-12-01; First posted 2016-07-13 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: functional tests — Test-retest reliability of physical function in hemodialysis patients

SUMMARY:
The investigators pretend to calculate values absolute and relative reliability that have not been yet reported (Short Physical Performance Battery, one-leg balance and Timed Up and go).

DETAILED DESCRIPTION:
Patients suffering from End Stage Renal Disease are commonly involved in haemodialysis treatment, which is the most common treatment at this stage. Haemodialysis substitutes the renal function but is associated with several alterations that lead to decrease in functional capacity and health related quality of life (HRQoL). Many studies show that functional capacity, physical activity level and HRQoL is significantly worse than their healthy sedentary age - matched counterparts. It is unknown if low physical activity, uraemia or anaemia are responsible for the decreased functional capacity of this cohort. Physical performance tests are frequently used to assess haemodialysis patients since is a feasible and low-cost evaluation. The purpose of the present study is quantified how the functional capacity changes over a -6 months period in a group of haemodialysis patients. Additionally the investigators pretend to calculate values absolute and relative reliability that have not been yet reported (Short Physical Performance Battery, one-leg balance and Timed Up and go).

ELIGIBILITY:
Inclusion Criteria:

* people under hemodialysis treatment at least 3 months
* be medicable stable
* complete all the physical tests

Exclusion Criteria:

* heart stroke in the previous 6 weeks of the study
* inferior limb amputation without artificial aids
* cerebral vascular disease (ictus, ischemic)
* disability to complete functional tests

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Chronic Kidney Diseases undergoing hemodialysis treatment
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2014-09; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery | It will perform the test twice with one to two weeks interval between the testing session
  Assess lower extremity, which includes objective performance-based measure of balance (side-by-side, semitanden and tandem), endurance (4m gait speed) and strength (five chair stands). Each component was scored from 0 to 4 and when summed yielded SPPB scores between 0 (poor) and 12 (best).

SECONDARY OUTCOMES:
One Leg Standing Test | It will perform the test twice with one to two weeks interval between the testing session
  Consist in maintain one leg stance for as long as possible. The test was considered normal if the one leg standing time reached 45 seconds.
Timed Up and Go | It will perform the test twice with one to two weeks interval between the testing session
  To stand up from a standard arms chair, walk 3 meters, turn back the cone walk back and sit down to the chair. The time in seconds is record.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Segura-Ortí, PhD, Principal Investigator — Professor at Universidad CEU Cardenal Herrera
Locations (1):
- Universidad CEU Cardenal Herrera, Moncada, Valencia, Spain

REFERENCES:
- [Background] Segura-Orti E, Martinez-Olmos FJ. Test-retest reliability and minimal detectable change scores for sit-to-stand-to-sit tests, the six-minute walk test, the one-leg heel-rise test, and handgrip strength in people undergoing hemodialysis. Phys Ther. 2011 Aug;91(8):1244-52. doi: 10.2522/ptj.20100141. Epub 2011 Jun 30. PMID 21719637